CLINICAL TRIAL: NCT01123980
Title: An Open-labelled, Randomised, Parallel Group, 3 Week run-in and 24 Week Treat-to-target Comparison of Biphasic Insulin Aspart 30 Once Daily Versus Insulin Glargine Once Daily Both in Combination With Metformin and Glimepiride in Chinese and Japanese Insulin Naive Subjects With Type 2 Diabetes
Brief Title: Comparison of the Blood Sugar Lowering Effect of Biphasic Insulin Aspart 30 and Insulin Glargine Both Combined With Metformin and Glimepiride in Chinese and Japanese Subjects With Type 2 Diabetes New to Insulin Treatment
Acronym: EasyMix
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-3756; U1111-1114-4112 (Other: WHO); JapicCTI-101139 (Other: JAPIC)
Record Dates: First submitted 2010-05-13; First posted 2010-05-14 (Estimated); Results first posted 2012-07-09 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70; Metformin; glimepiride; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BIAsp 30 (Experimental): 0.1-0.2 U/kg (starting dose) administered once daily (OD) immediately before dinner in combination with at least 1500 mg (Chinese patients) or 500 mg (Japanese patients) total daily dose of metformin and at least 4 mg glimepiride
  Interventions: Drug: biphasic insulin aspart 30; Drug: metformin; Drug: glimepiride
- Insulin glargine (Active Comparator): 0.1-0.2U/kg (starting dose) administered once daily (OD) at bedtime in combination with at least 1500 mg (Chinese patients) or 500 mg (Japanese patients) total daily dose of metformin and at least 4 mg glimepiride
  Interventions: Drug: metformin; Drug: glimepiride; Drug: insulin glargine

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — Treat-to-target titration according to titration algorithm. Subcutaneous (under the skin) injection once daily.
  Arms: BIAsp 30
Drug: metformin — China: Tablets, 500 mg. Min. 1500 mg/day.
  Japan: Tablets, 250 mg. Min 500 mg/day.
Drug: glimepiride — China: Tablets, 2 mg. Min. 4 mg/day.
  Japan: Tablets, 1 mg. Min. 4 mg/day.
Drug: insulin glargine — Treat-to-target titration according to titration algorithm. Subcutaneous (under the skin) injection once daily.
  Arms: Insulin glargine

SUMMARY:
This trial is conducted in Asia. The aim of this clinical trial is to investigate the blood sugar lowering effect of biphasic insulin aspart 30 once daily compared to insulin glargine once daily both in combination with metformin and glimepiride in Chinese and Japanese subjects with type 2 diabetes who have never received insulin before.

The trial is conducted as a phase 4 trial in China and phase 3 in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes treated with a maximum of three different types of oral anti-diabetic drugs (OADs) (including traditional Chinese medicine which contains active ingredients of known OADs) for more than 6 months
* Unchanged total daily dose of at least 1500 mg (Chinese patients) or 500 mg (Japanese patients) metformin for the last two months
* Unchanged total daily dose of at least half maximum recommended total daily dose of any insulin secretagogue for the last two months
* Insulin naive
* HbA1c between 7.0% and 10.0%
* FPG (fasting plasma glucose) equal to or above 6.1 mmol/L (110mg/dL)
* Body Mass Index (BMI) below 40.0 kg/m^2

Exclusion Criteria:

* Treatment with any thiazolidinedione (TZD) and GLP-1 (glucagon like peptide-1) receptor antagonists during the last 3 months before Visit 1 in this trial
* Any disease or condition which the Investigator feels would interfere with the trial
* Any contraindication to metformin or glimepiride (according to local labelling)

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 521 (Actual)
Dates: Start 2010-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (27):
- China (14):
  - Novo Nordisk Investigational Site, Beijing, Beijing Municipality
  - Novo Nordisk Investigational Site, Chongqing, Chongqing Municipality
  - Novo Nordisk Investigational Site, Fuzhou, Fujian
  - Novo Nordisk Investigational Site, Harbin, Heilongjiang
  - Novo Nordisk Investigational Site, Zhengzhou, Henan
  - Novo Nordisk Investigational Site, Nanjing, Jiangsu
  - Novo Nordisk Investigational Site, Wuxi, Jiangsu
  - Novo Nordisk Investigational Site, Nanchang, Jiangxi
  - Novo Nordisk Investigational Site, Dalian, Liaoning
  - Novo Nordisk Investigational Site, Shenyang, Liaoning
  - Novo Nordisk Investigational Site, Xi'an, Shaanxi
  - Novo Nordisk Investigational Site, Tianjin, Tianjin Municipality
  - Novo Nordisk Investigational Site, Shenyang
  - Novo Nordisk Investigational Site, Tianjin
- Japan (13):
  - Novo Nordisk Investigational Site, Asahikawa-shi, Hokkaido
  - Novo Nordisk Investigational Site, Chuo-ku, Tokyo
  - Novo Nordisk Investigational Site, Gifu City, Gifu
  - Novo Nordisk Investigational Site, Higashiku
  - Novo Nordisk Investigational Site, Kumamoto-shi,Kumamoto
  - Novo Nordisk Investigational Site, Minatoku
  - Novo Nordisk Investigational Site, Osaka
  - Novo Nordisk Investigational Site, Osaka-shi, Osaka
  - Novo Nordisk Investigational Site, Shimotsuka-gun
  - Novo Nordisk Investigational Site, Shimotsuke-shi, Tochigi
  - Novo Nordisk Investigational Site, Shizuoka
  - Novo Nordisk Investigational Site, Tagajō-shi
  - Novo Nordisk Investigational Site, Yokohama

REFERENCES:
- [Result] Yang W, Xu X, Liu X, Yang G, Seino Y, Andersen H, Jinnouchi H. Treat-to-target comparison between once daily biphasic insulin aspart 30 and insulin glargine in Chinese and Japanese insulin-naive subjects with type 2 diabetes. Curr Med Res Opin. 2013 Dec;29(12):1599-608. doi: 10.1185/03007995.2013.838155. Epub 2013 Sep 23. PMID 23998560
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 35 sites in two countries: China (21 sites) and Japan (14 sites).
Pre-assignment Details: At the screening, eligible subjects entered the run-in period before being randomised. During the 3 week run-in period, subjects switched from insulin secretagogue to glimepiride. During the last 2 weeks, the total dose of glimepiride was kept at 4mg/day. Subjects continued their pre-trial metformin dose.
Period: Overall Study
Arm/Group | BIAsp 30 | Insulin Glargine
Started | 261 | 260
Completed | 242 | 236
Not Completed | 19 | 24
Not completed — Adverse Event | 1 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Lost to Follow-up | 0 | 6
Not completed — Protocol Violation | 6 | 6
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Unclassified | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BIAsp 30 | Insulin Glargine | Total
Number analyzed (Participants) | 261 | 260 | 521
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (9.4) | 56.1 (9.9) | 56.3 (9.6)
Gender [Count of Participants; unit: Participants]
  Female | 114 | 119 | 233
  Male | 147 | 141 | 288
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 261 | 260 | 521
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 210 | 212 | 422
  Japan | 51 | 48 | 99
Height [Mean (Standard Deviation); unit: cm] | 165.3 (8.6) | 165.2 (8.2) | 165.3 (8.4)
Weight [Mean (Standard Deviation); unit: kg] | 70.0 (11.6) | 70.6 (12.5) | 70.3 (12.1)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.53 (3.39) | 25.76 (3.44) | 25.65 (3.41)
HbA1c (glycosylated haemoglobin) at randomisation [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.7 (0.88) | 8.14 (0.86) | 8.15 (0.87)
Duration of diabetes [Mean (Standard Deviation); unit: years] — Number of years since diagnosis
  years | 9.23 (7.15) | 9.47 (6.61) | 9.35 (6.88)
Diabetic complications at baseline [Number; unit: participants]
  Yes | 72 | 75 | 147
  No | 189 | 185 | 374

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Haemoglobin (HbA1c)
Time Frame: Week 0, week 24
Population: Full analysis set using LOCF (last observation carried forward) consists of all randomised subjects who were exposed to at least one dose of trial product(s)
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated haemoglobin
Arm/Group | BIAsp 30 | Insulin Glargine
Number analyzed (Participants) | 261 | 260
percentage of glycosylated haemoglobin | -0.68 (0.06) | -0.56 (0.06)
Statistical Analysis 1: Comparison: BIAsp 30 vs Insulin Glargine; H0: The mean treatment difference (BIAsp 30 minus insulin glargine) > 0.4%. HA: The mean treatment difference (BIAsp 30 minus insulin glargine) =< 0.4%. Sample size was calculated to achieve a power of at least 90%, assuming an equal change in HbA1c and a common standard deviation of 1.25%; Test type: Non-Inferiority or Equivalence — Non-inferiority was considered to be confirmed if the upper bound of the two-sided 95% confidence interval (CI) was below or equal to 0.4% or equivalent if the p-value for the one-sided test of H0: D > 0.4% against HA: D =< 0.4%, was less than or equal to 2.5%, where D is the mean treatment difference (investigational product minus comparator). Furthermore, superiority of BIAsp 30 OD over insulin glargine OD was shown if the upper limit of the 95% CI for the difference is lower than 0%; p < 0.001, ANCOVA — The p-values correspond to one-sided hypotheses of either non-inferiority or superiority, statistical significance level is 2.5%; The estimates are from a normal linear regression model with treatment, country and previous OADs as factors and baseline HbA1c as a covariate; Mean Difference (Net) = -0.12, 95% CI [-0.25 to 0.02], Standard Error of Mean 0.07

2. Secondary Outcome: 9-point Plasma Glucose Profiles
Description: Glycaemic control measured by 9-point plasma glucose (SPMG) profiles. The 9 timepoints for self-measurement during the day were: before breakfast, 2 hours after breakfast, before lunch, 2 hours after lunch, before dinner, 2 hours after dinner, before bedtime, at 2-4 a.m. and before breakfast the following day.
Time Frame: Week 24
Population: Full analysis set using LOCF (last observation carried forward) consists of all randomised subjects who were exposed to at least one dose of the trial product(s).
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | BIAsp 30 | Insulin Glargine
Number analyzed (Participants) | 261 | 260
mmol/L
  Before breakfast | 6.46 (0.09) | 6.49 (0.09)
  2 hours after breakfast | 10.18 (0.19) | 10.11 (0.19)
  Before lunch | 7.35 (0.17) | 7.22 (0.17)
  2 hours after lunch | 10.50 (0.20) | 10.22 (0.20)
  Before dinner | 7.67 (0.16) | 7.03 (0.16)
  2 hours after dinner | 9.36 (0.19) | 10.88 (0.19)
  Before bedtime | 8.14 (0.18) | 9.39 (0.18)
  At 2-4 a.m. | 6.58 (0.13) | 7.06 (0.13)
  Before breakfast the following day | 6.51 (0.10) | 6.35 (0.10)
Statistical Analysis 1: Comparison: BIAsp 30 vs Insulin Glargine; Repeated measures mixed model with an unstructured residual covarience matrix, including treatment, time, the treatment-by-time interaction, country and previous OADs as factors; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value for parallelism is overall test for parallel time profiles between treatment groups; Mean Difference (Final Values) = -0.03, 95% CI [-0.24 to 0.19] — Before breakfast
Statistical Analysis 2: Comparison: BIAsp 30 vs Insulin Glargine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value for parallelism is overall test for parallel time profiles between treatment groups; Mean Difference (Final Values) = 0.07, 95% CI [-0.45 to 0.58] — Two hours after breakfast
Statistical Analysis 3: Comparison: BIAsp 30 vs Insulin Glargine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value for parallelism is overall test for parallel time profiles between treatment groups; Mean Difference (Final Values) = 0.14, 95% CI [-0.31 to 0.58] — Before lunch
Statistical Analysis 4: Comparison: BIAsp 30 vs Insulin Glargine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value for parallelism is overall test for parallel time profiles between treatment groups; Mean Difference (Final Values) = 0.28, 95% CI [-0.26 to 0.82] — Two hours after lunch
Statistical Analysis 5: Comparison: BIAsp 30 vs Insulin Glargine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value for parallelism is overall test for parallel time profiles between treatment groups; Mean Difference (Final Values) = 0.64, 95% CI [0.22 to 1.06] — Before dinner
Statistical Analysis 6: Comparison: BIAsp 30 vs Insulin Glargine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value for parallelism is overall test for parallel time profiles between treatment groups; Mean Difference (Final Values) = -1.51, 95% CI [-2.03 to -1.00] — Two hours after dinner
Statistical Analysis 7: Comparison: BIAsp 30 vs Insulin Glargine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value for parallelism is overall test for parallel time profiles between treatment groups; Mean Difference (Final Values) = -1.25, 95% CI [-1.73 to -0.78] — Bedtime
Statistical Analysis 8: Comparison: BIAsp 30 vs Insulin Glargine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value for parallelism is overall test for parallel time profiles between treatment groups; Mean Difference (Final Values) = -0.47, 95% CI [-0.81 to -0.13] — 02 - 04 a.m
Statistical Analysis 9: Comparison: BIAsp 30 vs Insulin Glargine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value for parallelism is overall test for parallel time profiles between treatment groups; Mean Difference (Final Values) = 0.17, 95% CI [-0.06 to 0.40] — Before breakfast the following day

3. Secondary Outcome: Percentage of Subjects Achieving HbA1c Below 7.0%
Description: The percentage of subjects achieving the treatment target for glycosylated haemoglobin A1c after 24 weeks of treatment
Time Frame: Week 24
Population: as for outcome 2
Measure: Number; unit: percentage (%) of subjects
Arm/Group | BIAsp 30 | Insulin Glargine
Number analyzed (Participants) | 261 | 260
percentage (%) of subjects | 29.1 | 30.0
Statistical Analysis 1: Comparison: BIAsp 30 vs Insulin Glargine; The responder analysis was based on logistic regression model using treatment, country and previous OAD therapy (with or without a third OAD) as factors and baseline HbA1c as covariate; Test type: Superiority or Other; p = 0.8583, Regression, Logistic; Odds Ratio (OR) = 0.96, 95% CI [0.64 to 1.46] — The odds ratio and 95% confidence interval is for the HbA1c less than 7% treatment target were included

4. Secondary Outcome: Percentage of Subjects Achieving HbA1c Below or Equal to 6.5%
Description: The percentage of subjects achieving the treatment target for glycosylated haemoglobin A1c after 24 weeks of treatment
Time Frame: Week 24
Population: as for outcome 2
Measure: Number; unit: percentage (%) of subjects
Arm/Group | BIAsp 30 | Insulin Glargine
Number analyzed (Participants) | 261 | 260
percentage (%) of subjects | 14.9 | 14.2
Statistical Analysis 1: Comparison: BIAsp 30 vs Insulin Glargine; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.8013, Regression, Logistic; Odds Ratio (OR) = 1.07, 95% CI [0.64 to 1.79] — The odds ratio and 95% confidence interval is for the HbA1c below or equal to 6.5% treatment target were included

5. Secondary Outcome: Number of Hypoglycaemic Episodes - All
Time Frame: Weeks 0-24
Population: The safety analysis set contains all subjects exposed to at least one dose of investigational product(s).
Measure: Number; unit: episodes
Arm/Group | BIAsp 30 | Insulin Glargine
Number analyzed (Participants) | 261 | 260
episodes | 745 | 605

6. Secondary Outcome: Number of Hypoglycaemic Episodes - Severe and Minor
Description: Hypoglycaemic episodes (hypos) summarised based on American Diabetes Association classification (severe, documented symptomatic, asymptomatic, probable symptomatic, and relative hypoglycaemia) and according to additional definition (minor hypoglycaemia). Severe hypos: requiring another person to actively administer resuscitative actions. Minor hypos: symptoms with plasma glucose below 3.1 mmol/L (56 mg/dl), or any asympomatic plasma glucose below 3.1 mmol/L.
Time Frame: Weeks 0-24
Population: The safety analysis set contains all subjects exposed to at least one dose of investigational product(s).
Measure: Number; unit: episodes
Arm/Group | BIAsp 30 | Insulin Glargine
Number analyzed (Participants) | 261 | 260
episodes
  Severe | 0 | 1
  Minor | 154 | 125

7. Secondary Outcome: Number of Hypoglycaemic Episodes
Description: All episodes classified into nocturnal (time of onset between 00:00 (included) and 05:59 (included)).
Time Frame: Weeks 0-24
Population: The safety analysis set contains all subjects exposed to at least one dose of investigational product(s).
Measure: Number; unit: episodes
Arm/Group | BIAsp 30 | Insulin Glargine
Number analyzed (Participants) | 261 | 260
episodes | 97 | 63

ADVERSE EVENTS:
Time Frame: The adverse events were collected in a timespan of 24 weeks.
Description: The safety analysis set contains all subjects exposed to at least one dose of investigational products.
Arm/Group | BIAsp 30 | Insulin Glargine
Serious Adverse Events (participants affected / at risk) | 2/261 | 5/260
Other Adverse Events (participants affected / at risk) | 26/261 | 28/260
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIAsp 30 (N=261) | Insulin Glargine (N=260)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIAsp 30 (N=261) | Insulin Glargine (N=260)
Nasopharyngitis (Infections and infestations) | 26 (31) | 28 (37)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk reserves the right not to release data until specified milestones. This includes the right not to release interim results from clinical trials. At the end of the trial, one or more manuscripts for publication will be prepared in collaboration between Investigator(s) and Novo Nordisk. Novo Nordisk will not suppress or veto publications; however Novo Nordisk reserves the right to postpone publication and/or communication for a short time to protect intellectual property.